CLINICAL TRIAL: NCT00460980
Title: Effect of Virtual Reality Training by Novices on Laparoscopic Cholecystectomy in a Porcine Model
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: AAAB9401
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Gallstones
Keywords: resident training; laparoscopic skills; surgical skills assessment
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual reality laparoscopic simulator (Other): Virtual reality laparoscopic simulator training:
  Residents will participate in a structured approach to teaching laparoscopic skills to beginning surgeons with a virtual reality trainer will improve skills prior to actual operative experience.
  Interventions: Behavioral: Virtual reality laparoscopic simulator training

INTERVENTIONS:
Behavioral: Virtual reality laparoscopic simulator training — The aim of this project is to determine whether a structured approach to teaching laparoscopic skills to beginning surgeons with a virtual reality trainer will improve skills prior to actual operative experience. We aim to show that with the virtual reality trainer, operative skills will be improved and that overall operative time will be decreased.

SUMMARY:
This study proposes evaluation of an educational tool, a laparoscopic virtual reality simulator. The purpose of this study is to determine whether training on the LapSim Simulator transfers to improved laparoscopic cholecystectomy operative performance in an animal model.

DETAILED DESCRIPTION:
This is study protocol involves the training and evaluation of general surgery interns on a laparoscopic simulator (LapSim®, Surgical Science Ltd, Göteborg, Sweden, version 3.0.

ELIGIBILITY:
Inclusion Criteria:

* Surgical interns (PGY 1) are eligible
* Twenty-five (25) participants will comprise this group

Exclusion Criteria:

* Prior clinical experience with laparoscopic surgery as the assistant surgeon.
* Prior simulation training (mechanical, PC-based or otherwise).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Score on Global Outcomes Assessment of Laparoscopic Skills | 5 weeks, 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States